CLINICAL TRIAL: NCT01420302
Title: LOGIC-Insulin Computerized Algorithm-guided Versus Nurse-directed Blood Glucose Control in Critically Ill Patients: the LOGIC-1 Randomized Controlled Trial
Brief Title: LOGIC-Insulin Algorithm-guided Versus Nurse-directed Blood Glucose Control During Critical Illness
Acronym: LOGIC-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Greet Van den Berghe (Other)
Collaborators: Agency for Innovation by Science and Technology, Flanders, Belgium (Unknown); Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor-Investigator, Greet Van den Berghe, Head of Dept Intensive Care Medicine, KU Leuven
Organization: KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LOGIC-Insulin 1.1.1.; S 51956 (Other: University Hospitals Leuven); 80M0437 (Other: Belgian Federal Agency for Medicines and Health Products); ML 6079 (Other: IRB)
Record Dates: First submitted 2011-08-17; First posted 2011-08-19 (Estimated); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-04

CONDITIONS: Critical Illness
Keywords: critical illness; intensive care; insulin; glucose; algorithm; blood glucose control
MeSH Terms: conditions — Critical Illness; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Algorithm-guided versus Nurse directed Blood Glucose Control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LOGIC-Insulin (Experimental): Blood glucose control (80-110 mg/dL) guided by the LOGIC-Insulin algorithm
  Interventions: Procedure: LOGIC-Insulin
- Nurse-directed (Active Comparator): Nurse-directed blood glucose control (80-110 mg/dL)
  Interventions: Procedure: Nurse directed

INTERVENTIONS:
Procedure: Nurse directed — Nurse directed insulin titration to establish glycemic control in the target range of 80-110 mg/dL
  Other Names: Active comparator: titration-guidelines supported TGC
  Arms: Nurse-directed
Procedure: LOGIC-Insulin — Blood glucose control (80-110 mg/dL) guided by the LOGIC-Insulin algorithm
  Other Names: software guided TGC
  Arms: LOGIC-Insulin

SUMMARY:
The LOGIC-Insulin computerized software algorithm will be compared with a nurse-directed protocol, both targeting a blood glucose level of 80-110 mg/dL, in critically ill patients

DETAILED DESCRIPTION:
Critical illness typically causes elevated blood glucose concentrations, which have been associated with increased mortality. Strictly normalizing these blood glucose levels by intensive insulin therapy, called tight glycemic control, decreased morbidity and mortality in well-controlled single-center clinical studies. However, multi-center pragmatic trials failed to reproduce those effects, proving that the implementation of tight glycemic control in daily clinical practice is rather difficult.

A computerized algorithm, amongst others, may help the nurses in the titration of insulin to reach normal blood glucose levels and to avoid the particularly worrisome hypoglycemia.

The LOGIC-1 study is a single blinded randomized controlled trial. On admission patients will be randomly assigned to either tight glycemic control (80-110 mg/dL) by the computerized LOGIC-Insulin 3.0 algorithm or to tight glycemic control (80-110 mg/dL) by the nurse-directed protocol. Written informed consent will be asked from the patient in the case of elective surgery requiring post-operative ICU-admission. Proxy informed consent from the closest family member will be asked when the patient was admitted to the ICU in emergency. As blood glucose control by itself is essential in the management of critical illness, random allocation will be done on admission and written informed consent from the closest family member can be deferred to a maximum of 24 hours after randomization. The patient or family member can at all times withdraw from the trial without impact on his treatment. Allocation will be done in blocks (block size is unknown to the care givers responsible for treatment allocation), stratified into cardiac surgery and other reasons for ICU admission, by central computer randomization.

The time window for the study will be 14 days starting from admission to the ICU or when one of the following stop criteria will be met:

* Withdrawal of the informed consent
* Patient starts eating or drinking sugar containing liquids
* Patient is discharged from the ICU (including ICU deaths)
* Removal of arterial line or central venous line

Under the following conditions the study investigator/treating physician will be contacted and, if necessary, patients will be switched from LOGIC-Insulin to nurse-directed blood glucose control:

* Recurrent severe hypoglycemia (<40 mg/dL)
* Refractory hyperglycemia
* Any change in condition that compromises the safety of the patient, as judged by the investigator or treating physician

The common strategy for blood glucose control in both groups involves blood glucose measurements from arterial blood by a blood gas analyzer and the administration of insulin through a central line with a syringe pump.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more
* Admitted to the ICU
* Already receiving or needing insulin infusion for blood glucose control

Exclusion Criteria:

* Not critically ill (eating, not mechanically ventilated)
* Pregnant or breastfeeding
* Previous inclusion into the trial
* Included in other trial
* Moribund
* Diabetes coma
* No arterial line available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Mesotten, MD, PhD, Study Director — KU Leuven; Greet Van den Berghe, MD, PhD, Principal Investigator — KU Leuven; Tom Van Herpe, Eng, PhD, Principal Investigator — KU Leuven; Bart De Moor, Eng, PhD, Principal Investigator — KU Leuven
Locations (1):
- Dept Intensive Care Medicine, University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Van Herpe T, De Brabanter J, Beullens M, De Moor B, Van den Berghe G. Glycemic penalty index for adequately assessing and comparing different blood glucose control algorithms. Crit Care. 2008;12(1):R24. doi: 10.1186/cc6800. Epub 2008 Feb 26. PMID 18302732
- [Background] Van Herpe T, De Moor B, Van den Berghe G. Towards closed-loop glycaemic control. Best Pract Res Clin Anaesthesiol. 2009 Mar;23(1):69-80. doi: 10.1016/j.bpa.2008.07.003. PMID 19449617
- [Result] Van Herpe T, Mesotten D, Wouters PJ, Herbots J, Voets E, Buyens J, De Moor B, Van den Berghe G. LOGIC-insulin algorithm-guided versus nurse-directed blood glucose control during critical illness: the LOGIC-1 single-center, randomized, controlled clinical trial. Diabetes Care. 2013 Feb;36(2):188-94. doi: 10.2337/dc12-0584. Epub 2012 Sep 6. PMID 22961576
- See also: Leuven Laboratory Intensive Care Medicine — http://www.kuleuven.be/licm/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 22 August 2011 to 16 December 2011 in a 56-bed ICU of a tertiary referral university hospital
Period: Overall Study
Arm/Group | LOGIC-Insulin | Nurse-directed
Started | 149 | 151
Completed | 149 | 151
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LOGIC-Insulin | Nurse-directed | Total
Number analyzed (Participants) | 149 | 151 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (15) | 62 (14) | 63 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 58 | 119
  Male | 88 | 93 | 181
Region of Enrollment [Number; unit: participants]
  Belgium | 149 | 151 | 300
BMI (kg/m²) [Mean (Standard Deviation); unit: kg/m²] | 26.5 (5.5) | 25.9 (4.8) | 26.2 (5.2)
Apache II score (mean SD) [Mean (Standard Deviation); unit: units on a scale] — Acute Physiology and Chronic Health Evaluation (APACHE) II scores range from 0 to 71, with higher scores indicating a greater severity of illness
  units on a scale | 23 (10) | 24 (10) | 23 (11)
Admission type [Count of Participants; unit: Participants]
  After cardiac surgery | 76 | 74 | 150
  Transplantation | 19 | 25 | 44
  Medical | 26 | 23 | 49
  Other surgery | 28 | 29 | 57
Diabetes [Count of Participants; unit: Participants] | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Penalty Index (GPI) During the Intervention
Description: The GPI is an index (ranging from 0 to 100) derived from the blood glucose values that are outside the target level of 80-110 mg/dL, in both the hyperglycemic and the hypoglycemic ranges. The weight of the penalty score of a blood glucose measurement is proportional to the level of deviation from normoglycemia. The GPI is the average of all penalties that are individually assigned to all blood glucose values, based on an optimized smooth penalty function. Higher GPI scores indicate lower efficacy of glycemic control.
Time Frame: The GPI is the average of all penalties that are individually assigned to all blood glucose values obtained up to 14 days post-randomization, based on an optimized smooth penalty function.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | LOGIC-Insulin | Nurse-directed
Number analyzed (Participants) | 149 | 151
units on a scale | 9.8 [6.0 to 14.5] | 12.4 [8.2 to 18.5]
Statistical Analysis 1: Comparison: LOGIC-Insulin vs Nurse-directed; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Proportion of Patients With Severe Hypoglycemia (<40 mg/dL) During the Intervention
Description: Proportion of patients to have had one or more episodes of severe hypoglycemia (<40 mg/dL) during the intervention
Time Frame: up to 14 days post-randomization
Reporting Status: Not Posted

3. Secondary Outcome: Incidence of Severe Hypoglycemia (<40 mg/dL) During the Intervention
Description: Number of severe hypoglycemic values as a fraction of all blood glucose measurements during the intervention
Time Frame: up to 14 days post-randomization
Reporting Status: Not Posted

4. Secondary Outcome: Blood Glucose Level Per Treatment Group During the Intervention
Time Frame: up to 14 days post-randomization
Reporting Status: Not Posted

5. Secondary Outcome: Hyperglycemic Index (HGI) During the Intervention
Description: Adequacy of reaching and maintaining the target range for blood glucose during the intervention
Time Frame: up to 14 days post-randomization
Reporting Status: Not Posted

6. Secondary Outcome: Daily Maximal Blood Glucose Difference During the Intervention
Description: Marker of blood glucose variability
Time Frame: up to 14 days post-randomization
Reporting Status: Not Posted

7. Secondary Outcome: Proportion of Patients With Common Hypoglycemia (<60 mg/dL) During the Intervention
Description: Proportion of patients to have had one or more episodes of common hypoglycemia during the intervention
Time Frame: up to 14 days post-randomization
Reporting Status: Not Posted

8. Secondary Outcome: Interval Between Blood Glucose Measurements During the Intervention
Description: Marker of workload
Time Frame: up to 14 days post-randomization
Reporting Status: Not Posted

9. Secondary Outcome: Percentage of Time in Target Zone (80-110 mg/dL) During the Intervention
Description: Adequacy of reaching and maintaining the target range for blood glucose during the intervention
Time Frame: up to 14 days post-randomization
Reporting Status: Not Posted

10. Secondary Outcome: Length of Stay in ICU
Time Frame: up to 90 days post-randomization
Reporting Status: Not Posted

11. Secondary Outcome: Length of Stay in Hospital
Time Frame: up to 90 days post-randomization
Reporting Status: Not Posted

12. Secondary Outcome: Hospital Mortality
Description: Patients who will have been discharged from hospital before 90 days post-randomization will be regarded as survivors
Time Frame: up to 90 days post-randomization
Reporting Status: Not Posted

13. Secondary Outcome: Incidence of Common Hypoglycemia (<60 mg/dL) During the Intervention
Description: Number of common hypoglycemic values as a fraction of all blood glucose measurements during the intervention
Time Frame: up to 14 days post-randomization
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | LOGIC-Insulin | Nurse-directed
All-Cause Mortality (participants affected / at risk) | 19/149 | 10/151
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/151
Other Adverse Events (participants affected / at risk) | 0/149 | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes